CLINICAL TRIAL: NCT03724175
Title: The Role of Secondary Bile Acids in Intestinal Inflammation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Asst Prof-Med Ctr Line, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-47198
Record Dates: First submitted 2018-10-12; First posted 2018-10-30 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis; Pouchitis
Keywords: Ulcerative Colitis; Pouchitis
MeSH Terms: conditions — Colitis, Ulcerative; Pouchitis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ursodiol (ursodeoxycholic acid, UDCA) (Experimental): ursodiol (ursodeoxycholic acid, UDCA) 300 mg two times daily for 10 weeks to treat pouchitis in ulcerative colitis patients with antibiotic refractory or antibiotic dependent pouchitis
  Interventions: Drug: ursodiol (ursodeoxycholic acid, UDCA)

INTERVENTIONS:
Drug: ursodiol (ursodeoxycholic acid, UDCA) — ursodiol (ursodeoxycholic acid, UDCA) 300 mg two times daily for 10 weeks for UC pouchitis patients
  Other Names: NDC 0591-3159-01 Ursodiol Capsules, USP 300 mg

SUMMARY:
The cause of Inflammatory bowel disease (IBD) is unknown, but intestinal bacteria-involved in the production of molecules that impact health-are widely accepted to play a key role. A significant proportion of IBD patients with pouches (surgically created rectums after the diseased colon is removed) continue to have inflammation similar to their previous disease.

Only a few microbes are known to have the capability to modify primary bile acids (PBAs) made by the liver to secondary bile acids (SBAs). SBAs are some of the most common metabolites in the colon and play key roles in several diseases.

In this study the investigators will investigate if ursodeoxycholic acid (UDCA) may reduce inflammatory markers and improve quality of life (as assessed by validate survey) in those subjects with active antibiotic refractory or antibiotic dependent pouchitis.

DETAILED DESCRIPTION:
The cause of Inflammatory bowel disease (IBD) is unknown, but intestinal bacteria-involved in the production of molecules that impact health-are widely accepted to play a key role. A significant proportion of IBD patients with pouches (surgically created rectums after the diseased colon is removed) continue to have inflammation similar to their previous disease.

Only a few microbes are known to have the capability to modify primary bile acids (PBAs) made by the liver to secondary bile acids (SBAs). SBAs are some of the most common metabolites in the colon and play key roles in several diseases.

In previous study, the investigators examined bile acid levels in stool from pouches (surgically-created "rectums" made of small bowel) in colectomy-treated patients with ulcerative colitis (UC) versus colectomy-treated controls without inflammatory disease. This comparison revealed that certain SBAs are significantly decreased in stool from UC compared to control pouches.

In this study the investigators will investigate if ursodeoxycholic acid (UDCA) may reduce inflammatory markers and improve quality of life (as assessed by validate survey) in UC pouch patients (colectomy-treated patients with ulcerative colitis) with active antibiotic refractory or antibiotic dependent pouchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Male or female subjects, ≥18 years of age who have undergone an ileal pouch-anal anastomosis (IPAA) for UC.
3. History of pouchitis

   Documented evidence of active pouchitis, based on endoscopy, symptoms and histopathology, as follows:
4. Endoscopic score >=2 on the endoscopic component of a modified Mayo endoscopic score (where friability is scored as >2) Note: the area within 1 cm of the pouch staple, or pouch suture line, is not considered evaluable
5. Symptomatic disease (stool frequency):

   Subjects must demonstrate increased stool frequency compared to what is considered "normal" after their IPAA operation ("baseline"). Stool frequency must be an absolute value of > 6 stools per day, and > 3 stools per day above the post-IPAA "baseline". Note: The measurement of stool frequency will be a 7-day average rounded to the nearest integer. The most recent 7 days of data will be used to calculate the average.
6. Histology: evidence of disease.
7. Modified PDAI (mPDAI) score >= 5. The mPDAI consists of the symptom (range: 0-6) and endoscopy (range: 0-6) subscores.
8. Must have chronic antibiotic refractory or antibiotic dependent pouchitis.

Exclusion Criteria:

1. Lack of effective contraception Women of childbearing potential may not participate unless they are surgically sterile or are using adequate contraception.

   The following contraceptive methods are acceptable: hormonal (eg oral, injection, transdermal patch, implant, cervical ring), barrier (eg condom or diaphragm with spermicidal agent), intrauterine system or intrauterine device. If hormonal contraceptives are used by female subjects, they must be established for 6 weeks before the first administration of test product. Male sterilization is considered an acceptable form of contraception if the appropriate post-vasectomy documentation (absence of sperm) is provided in the subject's medical notes. Sexual abstinence is considered acceptable if this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (eg calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   Male subjects with female partners of child-bearing potential and female subjects who are neither surgically sterilized nor post-menopausal (defined as no menses for one year or a follicle-stimulating hormone value > 40 IU/L) will be required to use effective contraception throughout the study and for 30 days after.
2. Women who are pregnant or breastfeeding;
3. History of allergy or adverse event to UDCA;

   Stable use of concomitant medications for pouchitis is generally permitted, doses of concomitant medication, where taken, should be optimised in accordance with local/national practice guidelines, and dose levels and types of baseline medications for pouchitis will be documented and any changes during the study will be recorded. Changes in use of medications for pouchitis and high doses of oral steroids are not permitted. It is particularly important to maintain stable medication through to measurement of the primary end-point at Week 10. Criteria which would lead to exclusion of subjects from the study are described below:
4. Changes in dose to strong analgesia, such as opioid containing compounds within 4 weeks of the Screening Visit.
5. History of regular nonsteroidal anti-inflammatory drugs (NSAID) use.
6. Oral 5-aminosalicylate (5-ASA) compounds; exclude subjects who have discontinued or changed doses of oral 5-ASA within 4 weeks of the Screening Visit.
7. Oral budesonide > 6.0 mg/day is not permitted; exclude subjects who have received budesonide for < 6 weeks, or who have changed doses of budesonide within 4 weeks of the Screening Visit.
8. Oral steroids other than budesonide: exclude subjects who exceed a daily dose of 15 mg prednisolone or equivalent, who have received oral steroids for < 6 weeks, or who have changed dose within 4 weeks of the Screening Visit.
9. Use of rectal compounds is not permitted; these agents must be discontinued at the Screening Visit.
10. Immunosuppressant therapy (azathioprine, 6- mercaptopurine, methotrexate, cyclosporin); exclude subjects who have received treatment for < 12 weeks, or who have changed doses within 8 weeks of the Screening Visit.
11. Biological agents (Anti-tumour necrosis factor (anti - TNF) therapy, vedolizumab and / or ustekinumab); exclude subjects who have received biological agents for <6 months prior to the screening visit, or who changed doses of the biological agent within 6 months prior to the screening visit.
12. Previous use of UDCA is permitted: treatment course must have completed at least 12 weeks prior to the Screening Visit.
13. All other agents targeted to pouchitis, including experimental agents, must have been discontinued at least 8 weeks prior to the Screening Visit, or for a period equivalent to 5 half-lives (t1⁄2) of the agent (whichever is longer) It is acceptable to recruit subjects who remain on optimised, stable doses of oral 5-ASA, oral steroids (below the doses stipulated above) and immunosuppressants.

    It is acceptable to recruit subjects who terminated treatment with oral 5-ASA or oral steroids 4 weeks before the Screening Visit, or immunosuppressants 8 weeks before the Screening Visit.

    Note: Analgesic use should remain stable throughout the trial where possible. Paracetamol is the analgesic of choice.

    Note: VSL#3 probiotic treatment (and other probiotic treatments) will be permitted as long as maintained stable for 4 weeks prior to the Screening Visit, and maintained at a stable dose throughout the trial

    Also excluded are subjects with:
14. Anastomotic stricture
15. Unable to undertake endoscopic evaluation
16. Faecal incontinence due to anal sphincter dysfunction
17. Infections to cytomegalovirus or Clostridium Difficile
18. Faecal transplantation within 12 weeks of screening
19. Intestinal malabsorption
20. Pancreatic maldigestion
21. Suspected irritable pouch syndrome
22. Cuffitis (inflammation of the anal mucosa). Subjects with active antibiotic refractory pouchitis as the predominant condition, but who also have cuffitis, may be enrolled
23. Crohn's disease of the pouch; defined as either: a) complex perianal or pouch fistula and/or b) extensive pre-pouch ileitis with deep ulceration
24. Subjects with a history of neoplastic disease except for basal cell carcinoma or nonmetastatic squamous cell carcinoma of the skin
25. Subjects who are receiving or have received nasogastric/nasoenteric bottle feeding, an elemental diet, or total parenteral nutrition within the 2 weeks prior to Day 1
26. Subjects with a history of clinically significant and/or persistent haematologic, renal, hepatic, metabolic, psychiatric, central nervous system, pulmonary or cardiovascular disease; which in the investigator's opinion, would exclude entry into the study
27. Subjects with any laboratory tests considered clinically significant at screening
28. Subjects who may be unavailable for the duration of the trial, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason including, for example, inability to retain an enema formulation
29. Pelvic sepsis should be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve clinical response at week 10. | change from screening to end of treatment (10 weeks)
  Clinical response is defined as reduction of mPDAI score by >=2 points.

SECONDARY OUTCOMES:
Proportion of subjects who achieve remission at week 10. | change from screening at end of treatment (10 weeks)
  Remission is defined as mPDAI < 5 and reduction of mPDAI score by >=2 points.
Proportion of subjects who achieve endoscopic response at week 10. | change from screening at end of treatment (10 weeks)
  Endoscopic response is defined as reduction of modified MAYO (mMAYO)score by >=1 point.
Proportion of subjects who achieve endoscopic remission at week 10. | change from screening at end of treatment (10 weeks)
  Endoscopic remission is defined as mMAYO score <=1.
Proportion of subjects with a stool frequency represented by a Mayo subscore of <1 at Week 10. | change from screening at the end of treatment (10 weeks)
  Proportion of subjects with a stool frequency represented by a Mayo subscore of <1 at Week 10.
Mean change in Cleveland Global Quality of Life (CGQL) | change from screening, at week 6 and at end of treatment (10 weeks)
  Cleveland Global Quality of Life questionnaire (including current quality of life [0 being the worst and 10 being the best] ; current quality of health [0 being the worst and 10 being the best]; current energy level [0 being the worst and 10 being the best])
Mean change in erythrocyte sedimentation rate (ESR) | change from screening, at week 6 and at end of treatment (10 weeks)
  Mean change from baseline in erythrocyte sedimentation rate (ESR) at Week 6 and Week 10.
Mean change in C-reactive protein (CRP) | change from screening, at week 6 and at end of treatment (10 weeks)
  Mean change from baseline in C-reactive protein (CRP) at Week 10.
Mean change in fecal calprotectin | change from screening, at week 6 and at end of treatment (10 weeks)
  Mean change from baseline in fecal calprotectin at Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weingarden AR, Chen C, Zhang N, Graiziger CT, Dosa PI, Steer CJ, Shaughnessy MK, Johnson JR, Sadowsky MJ, Khoruts A. Ursodeoxycholic Acid Inhibits Clostridium difficile Spore Germination and Vegetative Growth, and Prevents the Recurrence of Ileal Pouchitis Associated With the Infection. J Clin Gastroenterol. 2016 Sep;50(8):624-30. doi: 10.1097/MCG.0000000000000427. PMID 26485102